CLINICAL TRIAL: NCT03795818
Title: An Open Clinical Trial of Interpersonal Psychotherapy for Adolescents With PTSD Symptoms
Brief Title: IPT-A for Adolescents With PTSD Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Laura Mufson, Professor of Medical Psychology (in Psychiatry), New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7717
Record Dates: First submitted 2018-12-24; First posted 2019-01-08 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Intervention Model Description: This is an open clinical trial of an psychosocial intervention for adolescents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IPT-A (Other): Interpersonal psychotherapy for adolescents (IPT-A) is a psychosocial treatment for adolescents. It has been shown to be effective for adolescents with depression. It is now being studied as to its benefit for adolescents who meet criteria for PTSD or have subthreshold PTSD symptoms.
  Interventions: Behavioral: Interpersonal Psychotherapy for Adolescents

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy for Adolescents — IPT-A is a psychosocial intervention for adolescents that focuses on improving interpersonal relationships that seem to be associated with the psychiatric symptoms.
  Other Names: IPT-A

SUMMARY:
In the present study, the investigators propose to 1) adapt Interpersonal Psychotherapy for Adolescents (IPT-A) as an intervention for adolescents who report elevated symptoms of posttraumatic stress disorder (PTSD) and/or meet Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria for PTSD; and 2) conduct a small open pilot study of IPT-A for PTSD. Ten adolescents ages 13 to 18 who meet DSM-5 criteria for a PTSD diagnosis or have elevated symptoms of PTSD (Child PTSD Symptom Scale [CPSS-5] ≥ 31) will be treated with 14-16 weeks of an adapted version of IPT-A. If participants have evidenced a decrease in PTSD symptoms (CPSS-5 < 31) they will also receive 3 months of once a month maintenance treatment and be assessed by a clinician evaluator at the conclusion of the 3 monthly sessions. If participants have not evidenced a decrease in PTSD symptoms (CPSS-5 ≥ 31), they will be referred for alternative treatments in the community and be assessed by a clinician evaluator 3 months following the completion of IPT-A. All evaluations and therapy sessions will be done over telehealth platform until able to be done in person.

DETAILED DESCRIPTION:
Please see the brief summary for study description.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents who meet criteria for DSM-5 diagnosis of PTSD or have elevated PTSD symptoms
2. English speaking adolescent and parent
3. Males and Females ages 13-18 years
4. Mild to moderate impairment in functioning

Exclusion Criteria:

1. Severe impairment in functioning
2. Diagnoses of substance abuse, Schizophrenia, Bipolar Disorder, Conduct Disorder, primary eating disorder, psychotic symptoms
3. Engagement in significant self-injurious behavior in the past 3 months
4. Active suicidality - presence of plan and/or intent
5. Intellectual disability or severe learning disability
6. Medical illness that may interfere with treatment
7. Current physical or sexual abuse
8. Open Administration for Children's Services (ACS) case
9. Currently receiving treatment for depression and/or PTSD or have begun a medication trial for another diagnosis within the previous three months

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Change in Child PTSD Symptom Scale (CPSS-5) | baseline, week 7, between weeks 14-16 (post-intervention), and at the 3 month follow-up, each time rating the 4 weeks prior to the assessment date.
  The Child Post-Traumatic Stress Disorder (PTSD) Symptom Scale (CPSS-5) is a self-report scale designed to assess PTSD symptoms in children and adolescents ages 8-18. The measure screens for stressful life events and asks about the emotional impact of these events in the 4 weeks prior to the assessment. Items are rated on a 5-point scale from 0 (not at all) to 4 (almost always) for how often the problem bothers the youth in the prior 4 weeks. A total symptom severity rating is calculated by summing the ratings of all 20 items and ranges from 0-80, with a higher score indicating greater symptom severity. The CPSS-5 will be used to assess change in PTSD symptoms through study completion at the 3-month follow-up assessment. The scale will be completed at baseline about the prior 4 weeks, at week 7 about the prior 4 weeks, between weeks 14-16 (post-intervention) about the prior 4 weeks, and at the 3-month follow-up assessment about the prior 4 weeks.
Change in Clinician-Administered PTSD Scale for DSM-5, Child/Adolescent Version (CAPS-CA-5) | baseline, between weeks 14-16 (post-intervention), and at the 3 month follow-up, each time rating the 4 weeks prior to the assessment date.
  The Clinician-Administered Post-Traumatic Stress Disorder (PTSD) Scale for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DMS-5) - Child/Adolescent Version (CAPS-CA-5) is a 30-item scale that assesses PTSD in children and adolescents ages 7 and older based on the 20 DSM-5 PTSD symptoms. Each item is given a severity rating based on symptom frequency and intensity. Ratings are given for the 4 weeks prior to each assessment timepoint. A total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms and ranges from 0-80, with a higher score indicating greater symptom severity. The CAPS-CA-5 will be used to assess change in symptoms through study completion at the 3-month follow-up assessment. The measure will be administered at baseline rating the prior 4 weeks, between weeks 14-16 (post-intervention) rating the prior 4 weeks, and at the 3-month follow-up assessment rating the prior 4 weeks.
Change in Clinical Global Scale of Illness - Improvement/Severity (CGI-I/S) | baseline, week 7, between weeks 14-16 (post-intervention), and at the 3 month follow-up, each time rating the 2 weeks prior to the assessment date
  The Clinical Global Scale of Illness - Improvement/Severity (CGI-I/S) is a 2-item clinician-rated instrument that assesses change in global illness severity and global improvement from baseline prior to treatment to study completion at the 3-month follow-up assessment. The improvement item is scored on a 7-point scale and ranges from 1 (very much improved since the initiation of treatment) to 7 (very much worse since the initiation of treatment). The severity item is scored on a 7-point scale and ranges from 1 (normal) to 7 (among the most extremely ill patients). It will be administered at baseline rating the prior 2 weeks, at week 7 rating the prior 2 weeks, between weeks 14-16 (post-intervention) rating the prior 2 weeks, and at the 3-month follow-up assessment rating the prior 2 weeks.

SECONDARY OUTCOMES:
Change in Mood and Feelings Questionnaire (MFQ) | baseline, week 7, between weeks 14-16 (post-intervention), and at the 3 month follow-up, each time rating the 2 weeks prior to the assessment date
  The Mood and Feelings Questionnaire (MFQ) is a 33-item self-report measure completed by the parent and adolescent to identify symptoms of depression in children and adolescents ages 6-17. Items are scored from 0 (not true) to 2 (true). A total score is calculated by summing the point values of all items and ranges from 0 to 66, with higher scores indicating more severe depressive symptoms. The measure will be completed at baseline about the prior 2 weeks, at week 7 about the prior 2 weeks, between weeks 14-16 (post-intervention) about the prior 2 weeks, and at the 3-month follow-up assessment about the prior 2 weeks. Scores at these timepoints will enable assessment of change in symptoms through completion of the study at the 3-month follow-up assessment.
Change in Social Adjustment Scale-Self Report (SAS-SR) | baseline, week 7, between weeks 14-16 (post-intervention), and at the 3 month follow-up, each time rating the 2 weeks prior to the assessment date
  The Social Adjustment Scale-Self Report (SAS-SR) is a 23-item scale that assesses social adjustment/functioning for the past 2 weeks in 5 areas: overall adjustment, school behavior, relationships with friends, relationships with family, and dating. Items are scored on a Likert scale from 1 to 5. A total score is calculated by averaging all items. Subscale scores are calculated by averaging all items within each subscale. The total and subscale scores range from 1-5, with higher scores indicating more impaired social adjustment. The SAS-SR will be completed at baseline about the prior 2 weeks, at week 7 about the prior 2 weeks, between weeks 14-16 (post-intervention) about the prior 2 weeks, and at the 3-month follow-up assessment about the prior 2 weeks. Ratings will provide information regarding change in social adjustment through study completion at the 3-month follow-up assessment.
Change in Columbia-Suicide Severity Rating Scale (C-SSRS) | lifetime from birth to baseline time period, the month (4 weeks) prior to the initial baseline assessement prior to treatment, and at weeks 7, 14-16 (post intervention) and 3 month follow-up ratings on behavior since prior assessment up to 36 weeks.
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinician-administered measure that collects information on suicidal behavior, suicide attempts, and presence and intensity of suicidal ideation. The majority of the items are scored as yes or no for being present, severity items for suicidal ideation are scored regarding frequency and intensity. A numerical Suicidal Ideation Score is equivalent to the maximum category of items 1-5 that is present at the assessment, where 0 is no suicidal ideation and 5 is active suicidal ideation with specific plan or intent. The baseline version will assess lifetime of the adolescent and past 4 weeks of suicidal ideation and behavior. At week 7, between 14-16 weeks (post-intervention), and at the 3-month follow-up timepoint, it will be administered and assess suicidal ideation and behavior for the past 7 weeks at weeks 7 and 14-16 (post-intervention), and the past 36 weeks at the 3-month follow-up assessment.
Change in Children's Global Assessment Scale (CGAS) | baseline, week 7, between weeks 14-16 (post-intervention), and at the 3 month follow-up, each time rating the past 4 weeks prior to the assessment date
  The Children's Global Assessment Scale (CGAS) is a clinician-rated scale that assesses overall/global impairment across aspects of the child's life for the 4 weeks prior to the assessment. It has been found to be a reliable instrument for assessing impairment in children with psychiatric disorders. Based on clinical interview, the evaluator assigns a single score for the person's level of impairment in various domains of his/her life including relationships, school, work, and symptomatology in the 4 weeks prior to the assessment. A single global rating is provided on a scale of 1-100, with 100 being no impairment. It will be completed at baseline, week 7, between weeks 14-16 (post-intervention), and at the 3-month follow-up assessment, rating the 4 weeks prior to each of these timepoints. The repeated timepoints will allow assessment of change from baseline through the study completion at the 3-month follow-up assessment.
Change in Conflict Behavior Questionnaire (CBQ) | baseline, week 7, between weeks 14-16(post-intervention), and at the 3 month follow-up, each time rating the past 2 weeks prior to the assessment date.
  The Conflict Behavior Questionnaire is a self-report that assesses the parent-child relationship for the 2 weeks prior to the assessment. It has been found to be a reliable measure of the quality of the relationship between mother and adolescent and father and adolescent. It is completed both by the adolescent about the parents and the parent about the adolescent. It is a 20-item scale scored on a true/false scale. The total score is calculated by summing the point values of all of the items and ranges from 0-20. Higher scores indicate greater conflict in the relationship. The CBQ will be completed at baseline, week 7, between weeks 14-16 (post-intervention), and at the 3-month follow-up assessment, rating the 2 weeks prior to each of these timepoints. The repeated timepoints will allow assessment of the change from baseline through the study completion at 3-month follow-up assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mufson, Ph.D., Principal Investigator — Columbia University/NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No